CLINICAL TRIAL: NCT05053672
Title: The Respiratory Therapy Method Based on Short-term Intermittent Exposures Hypoxia and Hyperoxia (ReOxy Therapy) in the Rehabilitation of Chronic Low Back Pain Patients With Cardiac or Pulmonary Comorbidities: a Randomized Controlled Trial
Brief Title: ReOxy Therapy in the Rehabilitation of Chronic Low Back Pain Patients With Comorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4 11052021
Record Dates: First submitted 2021-08-26; First posted 2021-09-22 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
Keywords: low back pain; chronic lumbar back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective analysis in a 3-arm, randomized single-blind and placebo controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional therapy back pain treatment (No Intervention): Participants randomized to сonventional therapy group will receive complex rehabilitation program including physical exercise, phonophoresis with hydrocortisone, lumbar region massage, acupuncture within 2 weeks.
- Conventional physiotherapy therapy back pain treatment + ReOxy-therapy (Active Comparator): Participants randomized to Active Comparator group will receive complex rehabilitation program and 10 ReOxy-therapy sessions within 2 weeks (5 sessions per week).
  Interventions: Device: ReOxy
- Conventional physiotherapy therapy + Sham ReOxy-therapy (Placebo Comparator): Participants randomized to Placebo Comparator group will receive complex rehabilitation program and 10 sham ReOxy-therapy sessions within 2 weeks (5 sessions per week).
  Interventions: Device: Sham ReOxy

INTERVENTIONS:
Device: ReOxy — ReOxy therapy is a protocol which employs passive (the patient is at rest), short (up to 10 min) mild normobaric hypoxic exposures alternated with similar duration intervals of breathing hyperoxia (up to 5 min). The gas mixtures are supplied to a patient via facial mask on continued measuring of oxygenation status of the patients, lasting about 45 min in total per treatment session.
  The hypoxic load will be individually adjusted, based on the results of a preliminary hypoxic test. The patient inhales air with low oxygen content (10-14%) at atmospheric pressure in a continuous mode through a mask withing 10-min.
  During the ReOxy - treatment session, the software automatically adjusts the gas mixture switching, based on changes in physiological parameters (blood oxygen saturation and heart rate) in response to hypoxic and hyperoxic impact (biofeedback control).
  Arms: Conventional physiotherapy therapy back pain treatment + ReOxy-therapy
Device: Sham ReOxy — Placebo treatment with 'sham' ambient air breathing to simulate ReOxy-therapy sessions. Placebo-mode breathing set visually similar to standard breathing set but have a mask with open intake valve. The masks are chosen in a way to provide maximum degree of similarity to reduce the risk of unblinding on the patient-side.
  Arms: Conventional physiotherapy therapy + Sham ReOxy-therapy

SUMMARY:
The aim of this study is to assess the effect of the respiratory therapy method based on short-term intermittent exposures to hypoxia and hyperoxia (ReOxy therapy) on the pain intensity, restoration of the lumbar range of motion, physical capacity, disability, mental and vegetative status in Chronic Low Back Pain patients with Multiple Chronic Conditions.

DETAILED DESCRIPTION:
This is a randomized, single-blinded, placebo-controlled trial, with chronic non-specific low back pain with multiple chronic conditions. Comorbidity constitutes a serious challenge for rehabilitative medicine - significantly reduces the patients' quality of life and restoration of the working capacity.

The objective of the present study will be to evaluate the effectiveness of the combined non-medicinal rehabilitation programe which include a course of ReOxy- therapy and conventional therapy back pain treatment.

90 patients will be randomly allocated to three treatment groups: experimental ("hypoxic group" - ReOxy therapy + conventional therapy back pain treatment), placebo ("sham hypoxic group"- sham- ReOxy therapy + conventional therapy back pain treatment) and control (only conventional therapy back pain treatment).

The clinical outcomes will be obtained at the completion of treatment (2 weeks) and at 1 month after randomization. The statistical analysis will follow the intention-to-treat principles and the between-group differences will be calculated by using mixed linear models.

The outcomes of interest are pain intensity, lumbar range of motion function, general physical and mental status.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-specific chronic low back pain for at least 3 months;
* A pain intensity of at least 5 points measured by 0 -10 points pain rating scale;
* Co-morbidity - IHD and/or CHF and/or COPD and/or chronic bronchitis)
* Willing and able to consent, complete all assessment and study procedures;

Exclusion Criteria:

* Specific types of back pain (metastatic cancer or bone cancer or secondary cancers, vertebral fractures, spinal infection, active inflammatory disease);
* Low back surgery within past 3 months;
* Serious cardiovascular, cerebrovascular, neuromuscular and other systemic diseases or other diseases affecting physical activity;
* Any significant systemic illness or medical condition that could affect safety or compliance with study;
* Major active or chronic unstable psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year;
* Tumour disease except being successfully treated and off treatment with >2 years. Tumour disease except being successfully treated and off treatment with >2 years.
* Use of other investigational agents or interventions one month prior to entry and for the duration of the trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Back pain intensity will be measured by the Visual Analog Scale | Baseline, end of the 2-nd week
  Visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. The VAS consists of a 10cm horizontal line with the words "no pain" and "worst pain" at the line's end. VAS is a reliable and valid tool to reliable and valid tool to measure pain intensity measure pain intensity.

SECONDARY OUTCOMES:
Back pain intensity | Baseline and 1-month post randomization
  Back pain intensity will be measured by the Visual Analog Scale Visual analogue scale (VAS) is a simple and frequently used method for the assessment of variations in intensity of pain. The VAS consists of a 10cm horizontal line with the words "no pain" and "worst pain" at the line's end. VAS is a reliable and valid tool to reliable and valid tool to measure pain intensity measure pain intensity.
Roland Disability Questionnaire (RDQ) | Baseline and 1-month post randomization
  The Roland-Morris Questionnaire is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale
Lumbar Range of Motion | Baseline, end of the 2-nd week
  Will be evaluated through the finger-to-floor test. Participant try to reach the floor with his fingertip by bending forward in the same time knees are kept extended. The distance between fingertips and floor are measured in centimetres by examiner.
Change of lower back flexibility | Baseline, end of the 2-nd week
  Will be evaluated through Schober test (positive/negative). The examiner places one finger 5cm below the mark pproximately at the level of L5 and another finger at about 10cm above this mark. The patient is then instructed to touch his toes. If the increase in distance between the two fingers on the patients spine is less than 5cm then this is indicative of a limitation of lumbar flexion.
6 min-walking test distance | Baseline, end of the 2-nd week
  Change in walking distance in meters during a 6-min period over a corridor of 30m length
Hospital Anxiety and Depression Scale, HADS | Baseline and 1-month post randomization
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3. The scale is devided into 2 parts: (1) anxiety (minimum score 0, maximum sore 21) and (2) depression (minimum score 0, maximum sore 21).
  Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
Bergen Insomnia Scale (BIS) | Baseline and 1-month post randomization
  The BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IV-TR (American Psychiatric Association). Higher values indicate higher levels of insomnia severity.

OTHER OUTCOMES:
HR recovery after the 6-minute walk test | Baseline and end of the 2-nd week
  HR recovery measured by sphygmomanometer after the 6-minute walk test
SAD/DAD recovery after the 6-minute walk test | Baseline and end of the 2-nd week
  SAD/DAD recovery measured by sphygmomanometer after the 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Nadezhda Lyamina, M.D., Principal Investigator — Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine
Locations (1):
- Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine, Dept. No. 9, Moscow, Russia